CLINICAL TRIAL: NCT02688673
Title: Safety and Therapeutic Efficacy of DC Vaccine Combined With Cytokine-induced Killer Cells in Patients With Extensive-Stage Small- Cell Lung Cancer: a Phase I/II Study
Brief Title: DC Vaccine Combined With CIK Cells in Patients With SCLC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Affiliated Hospital to Academy of Military Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 307-DC/CIK-SCLC
Record Dates: First submitted 2016-02-18; First posted 2016-02-23 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2015-10

CONDITIONS: Small- Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: adenovirus-transfected autologous DC vaccine plus CIK cells

SUMMARY:
The aim of this study is to evaluate the safety and efficacy of dendritic cells (DC) combined with cytokine-induced killer (CIK) cells treatment patients with Extensive-Stage Small-Cell Lung Cancer. Experimental adopted recombinant adenovirus-code MUC1 and Survivin transfected DC, which are used for DC-based immunotherapy. Based on the results of our previously preclinical research with DC combined with CIK cells, the investigators plan to perform the clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed diagnosis of Small- Cell Lung Cancer
* Age >18 years at time of consent
* Received standardized treatment of Small-Cell Lung Cancer
* Interval between the last standardized treatment and DC/CIK treatment ≥ 4weeks
* KPS (Karnofsky performance scale) >60
* Patient's written informed consent
* No severe viral or bacterial infections
* Predicted survival >3 months

Exclusion Criteria:

* Clinically relevant diseases or infections (HBV, HCV, HIV)
* Females who are pregnant or nursing
* Immunosuppressant treatment
* Currently participating in another clinical trial
* Unfit for participating in this clinical trial in investigators' opinions

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-08 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
objective rate response (CR+PR) as measured by RECIST criteria | 4 weeks after DC/CIK treatment]

SECONDARY OUTCOMES:
number of participants with adverse events | 3 days within DC/CIK treatment